CLINICAL TRIAL: NCT07134192
Title: Fluorescence-Guided Optimization of Sarcoma Margins
Acronym: FOCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113942; 1-10-72-34-25 (Other: Scientific Ethics Committees for the Central Denmark Region)
Record Dates: First submitted 2025-08-13; First posted 2025-08-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Sarcoma of the Trunk and Extremities; Sarcoma
Keywords: Sarcoma; ICG; Indocyanine green; Fluorescence Guided Surgery; FGS; STS; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: National multicenter interventional cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorescence-guided surgery cohort (Experimental): Patients with intermediate-to-high grade sarcomas eligible for curative surgical treatment at time of surgery. Surgery will be augmented by guidance through the use of a near-infrared camera and fluorescent dye administered the day prior to surgery.
  Interventions: Procedure: Fluorescent-guided Surgery

INTERVENTIONS:
Procedure: Fluorescent-guided Surgery — Surgical treatment of the patient group will include the administration of a fluorescent dye and intraoperatively the resection will be aided and guided by the fluorescent signal. The wound bed will be inspected, areas with fluorescent signal will be excised and obtained separately for histopathology. Patients will receive the current post-operative standard of care for sarcoma patients

SUMMARY:
This is a Danish national multicenter prospective cohort study to evaluate if fluorescence-guided surgery (FGS) using indocyanine green (ICG) can reduce the rate of positive margins following sarcoma resection.

DETAILED DESCRIPTION:
This is a Danish national multicenter prospective cohort study to evaluate if fluorescence-guided surgery (FGS) using indocyanine green (ICG) can reduce the rate of positive margins following sarcoma resection.

Biopsy verified intermediate-to-high grade sarcoma of the extremity or trunk wall are eligible for inclusion. To be included there must be curative intent at time of surgery.

The primary endpoint will be re-resection within 30 days due to positive margins on the initial resection. Tumor characteristics and margin status from pathology reports will be recorded. Data on reoperations due to other factors, positive margins without planned reoperation, or death will also be collected. Participants will undergo surgery with ICG administered and guided using the SPY-PHI.

The prospective cohort will be compared to a historic cohort having received standard of care treatment. The historic cohort is included to act as a control group to compare with the new procedure. The data is derived from the Danish Sarcoma Database and permissions for this is in process. This data does not involve access to patient EMRs.

Patients will receive an intravenous bolus of 1 mg/kg fluorescent ICG dye 16-24 hours before surgery. During surgery, consecutive measurements will be recorded using the SPY-PHI. Surgical resection will be guided by the fluorescent signal. The wound bed will be inspected, areas with fluorescent signal will be excised and obtained separately for histopathology. Patients will receive the current post-operative standard of care for sarcoma patients.

Approximately 20 minutes of additional surgical time is expected.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy verified intermediate-to-high grade sarcoma of theextremity or trunk wall
* Age>18 years old
* Tumor operable
* Curative intent at time of surgery
* Consent of patient

Exclusion Criteria:

* History of allergic reaction to iodine-containing pharmaceuticals
* End-stage renal disease or eGFR <15
* Patient decision
* Lack of capacity
* Inoperability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Reresection | 30 days
  Reresection within 30 days will be used as primary endpoint as a proxy for histopathologically positive margin status following surgery which would require reoperation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Baad-Hansen, MD, PhD, Study Director — Orthopedic Surgical Department, Aarhus University Hospital; Christian Kveller, MD, Principal Investigator — Orthopedic Surgical Department, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No